CLINICAL TRIAL: NCT00455286
Title: High-Dose Methotrexate Plus Steroid Followed by Concurrent Whole Brain Chemoradiation With Temozolomide for Immunocompetent Patients With Primary Central Nervous System Lymphoma - a Phase II Study
Brief Title: a Phase II Study in Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Taichung Veterans General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1406
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: CNS Lymphoma
MeSH Terms: interventions — Methotrexate; Methylprednisolone; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methotrexate
Drug: Methylprednisolone
Drug: Temozolomide

SUMMARY:
In this study we will test the hypothesis that concurrent chemoradiation (CCRT) with temozolomide after induction chemotherapy by conventional high-dose methotrexate (HD-MTX) plus dexamethasone may be an effective and well tolerated treatment for immunocompetent patients with PCSNL. Corticosteroid can effectively reduce brain edema and corticosteroid alone has resulted in complete or partial remission in about 40% patients with PCNSL. To enhance local disease control, CCRT with temozolomide will be used in the study. Temozolomide is a well-tolerated oral alkylating agent that is able to permeate the BBB. Concurrent temozolomide with WBRT has shown superior effect to WBRT alone for the treatment of metastatic brain tumors and glioblastoma multiforme. In addition, temozolomide has single-agent activity for PCNSL (21% CR in relapsed or refractory PCNSL in a phase II trial).

This is an open-label, non-randomized, multi-center phase II study. The primary end point of is the complete response rate. This study is a two-stage design for testing non-inferiority of the proposed treatment as compared to the approximately 80% response rate reported for conventional treatment. Assuming a non-inferiority margin of 20%, a sample size of 25 subjects, which provides an 80% power for establishment of non-inferiority. At the first stage, 15 subjects are to be enrolled. If equal to or more than 6 patients achieve complete response, the study would accrue additional 10 subjects. The treatment regimen is as follows.

Induction chemotherapy: MS regimen (repeated every 14 days, total 4 cycles)

* Methotrexate 3.5 g/m2 i.v. infusion 4 hours on day1
* Methylprednisolone 200 mg/m2/day i.v. infusion 30 minutes, on day1-4 Concurrent chemoradiotherapy (CCRT)
* Whole brain radiation therapy (WBRT) 2 Gy per fraction daily, 5 days per week Temozolomide 75 mg/m2/day orally daily, only on the days of WBRT

DETAILED DESCRIPTION:
5 PATIENT SELECTION 5.1 Eligibility Criteria

Patients must fulfill all the following criteria to be eligible for admission for the study:

1. Histologically proven central nervous system lymphoma of brain parenchyma with or without leptomeningeal involvement.
2. No evidence of systemic lymphoma.
3. Age between 18 years and 75 years.
4. With at least one measurable lesion, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 10 mm. See Section 10.2.1 for the evaluation of measurable disease.
5. Laboratory requirements :

   * Hematology: Neutrophils≧ 1500/mm3, Hemoglobin≧ 10 g/dL, and Platelet count≧ 100000/mm3.
   * Hepatic function: Total bilirubin level≦ 1.5x upper normal limit (UNL), ALT (SGPT) and AST (SGOT)≦ 2.5 x UNL.
   * Renal function: Creatinine≦ 1.5 mg/dL.
6. No prior malignancy (excluding in situ carcinoma of the cervix or non- melanomatous skin cancer) unless disease free for at least 5 years.
7. Signed informed consent.
8. Patients must be accessible for treatment and follow-up. 5.2 Ineligibility Criteria Patient meets any of the following will be excluded form the study.

<!-- -->

1. Patients who are seropositive for HIV, AIDS, use of immunosuppressant or who are post organ transplant are not eligible.
2. Previously treated with chemotherapy, radiotherapy or other investigational agents. Patients with corticosteroid use are considered eligible.
3. With ocular involvement or with any lesion beyond brain parenchyma except leptomeningeal.
4. Pregnant, or lactating patients; patients of childbearing potential must implement adequate contractive measures during study participation.
5. Other serious illness or medical conditions:

   * Congestive heart failure or unstable angina pectoris. High risk uncontrolled arrhythmias.
   * Uncontrolled infection (active serous infections that are not controlled by antibiotics.
6. Concurrent treatment with any other experimental drugs.

6 PLAN OF THE STUDY 6.1 Study Design This is an open-label, multi-center phase II study designed to access the response rate (including CR, CRu and PR, definition refers to 10.2.2) in patients with primary central nervous system lymphoma receiving MS followed by CCRT with temozolomide. The secondary objectives are to access time to progression and to the safety of the combination in this patient population.

6.2 Sample Size The primary end point of this phase II study is the objective tumor response rate. This study is a two-stage design for testing non-inferiority of the proposed treatment as compared to the approximately 80% response rate reported for conventional treatment. Assuming a non-inferiority margin of 20%, a sample size of 25 subjects, which provides an 80% power for establishment of non-inferiority, was selected based on the method described in Batchelor et al.7 At the first stage, 15 subjects are to be enrolled. If fewer than six patients respond (the one-sided 93% upper bound of the observed response rate is lower than 60%), the study would be terminated. Otherwise, the study would accrue additional 10 subjects. At the end of second stage, if the one-sided lower 95% confidence limit of the point estimate of the response rate is greater than or equal to 60%, the hypothesis that the study treatment is inferior to the conventional treatment would not be rejected.

7.2 Treatments Schedules

* Patient who meet the inclusion and exclusion criteria will receive induction chemotherapy (MS regimen).
* If patient with leptomeningeal involvement or CSF+ at diagnosis, intrathecal methotrexate will be given during the period of induction chemotherapy.
* Two to 4 weeks after completion of induction chemotherapy, if the disease is confined within brain parenchyma or completely remitted, concurrent temozolomide with whole brain radiation will be started. (Table 1. is and example of 2 weeks after induction chemotherapy).
* If the disease is beyond brain parenchyma or persistent leptomeningeal involvement during or after completion of induction chemotherapy, the patient should be taken off the study.

7.3 Induction Chemotherapy (MS regimen)

* Methotrexate 3.5 g/m2 i.v. infusion 4 hours on day1
* Methylprednisolone 200 mg/m2/day i.v. infusion 30 minutes, on day1-4

  1. Cycles will be repeated every 2 weeks on week 1, 3, 5, and 7, if no evidence of disease progression.
  2. Sample orders are detailed in Appendix V.
  3. Hydration and urine alkalization: It is mandatory that all patients receive adequate hydration and urine alkalization (keep urine pH >7) post the methotrexate infusion.
  4. Antiemetics: All patients could receive prophylactic antiemetic medication 30 minutes before each methotrexate infusion. 5-HT3 antagonists are recommended.
  5. Leucovorin rescue: Leucovorin 30 mg i.v. every 6 hours should be started since 24 hours after the start of methotrexate infusion until serum methotrexate level is less than 0.05 mcM and at least 8 doses.

     * In patients with delayed early methotrexate elimination and/or evidence of acute renal injury (serum methotrexate level of 50 mcM or more at 24 hours, or 5 mcM or more at 48 hours after administration, or serum creatinine≧ 2.0 mg/dL at 24 hours) give leucovorin 150 mg IV every 3 hours until methotrexate level is less than 1 mcM then 30 mg IV every 6 hours until methotrexate level is less than 0.05 mcM.
     * In patients with delayed late methotrexate elimination (serum methotrexate level remaining above 0.2 mcM at 72 hours or more than 0.05 mcM at 96 hours after administration), continue leucovorin 30 mg i.v. every 6 hours until methotrexate level is less than 0.05 mcM;
  6. Others: Allopurinol and antacid are recommended during the first 5 days of each cycle.

7.4 Intrathecal Methotrexate  Methotrexate 12 mg intrathecal injection on day 8 of induction chemotherapy

1. Only for leptomeningeal involvement or CSF cytology positive.
2. Cycles repeat every 2 weeks on week 2, 4, 6, and 8, if no evidence of disease progression. If the induction chemotherapy with MS is delayed, intrathecal methotrexate schedule will be decided by treating physician.
3. If CSF+ is newly found during treatment, the patient must be off protocol.
4. Leucovorin 15 mg p.o. bid should be used 24 hours after intrathecal methotrexate for 3 days.

7.5 Concurrent Whole Brain Radiation with Temozolomide 7.5.1 Whole Brain Radiation Therapy

* Whole brain radiation therapy (WBRT) 2 Gy per fraction daily, 5 days per week

  1. For patients with CR or CRu after induction chemotherapy, a total of 30 Gy will be given; for patients with non-CR/ CRu after induction chemotherapy, a total of 36 Gy will be given.
  2. WBRT should be initiated within 2-4 weeks after starting the last induction chemotherapy if no active infection or life threatening complication is noted.
  3. Continuation of WBRT as schedule is suggested unless the treating physicians judge the patient's condition to be inappropriate to receive WBRT.
  4. Physical Factors: Treatment will be delivered using megavoltage machines with photon beams ranging from 4 to 8 MV. The minimum dose rate at the midplane in the brain on the central axis must be 0.50 Gy/minute. Electron, particle, or implant therapy is not permissible.
  5. Simulation, Immobilization, Localization: The patient will be treated in the supine position. Adequate immobilization and reproducibility of position are encouraged. The target volume will cover the brain and the meninges to the foramen magnum.
  6. Treatment Planning: Treatments must be delivered through parallel opposed or 5 degree RAO-LAO fields that cover the entire cranial contents. There should be beam fall-off of at least 1 cm. The eyes will be excluded from the beam either by field arrangement or shielding.
  7. Stereotactic radiosurgery and intensity modulated radiotherapy (IMRT) are not allowed.

     7.5.2 Temozolomide
* Temozolomide 75 mg/m2/day orally daily, only on the days of WBRT

  1. Criteria for starting Temozolomide: The initiation of temozolomide will be based upon complete blood counts (CBC) obtained within 48 hours prior to starting the treatment. If ANC is ≥ 1,000/mm3 and platelet count is ≥ 75,000/mm3, the temozolomide may be started. If study drug cannot be administered on the scheduled day of dosing, the CBC will be repeated every 3 days.
  2. Since capsules of study drug are available in 20 and 100 mg capsules in Taiwan, all doses will be rounded up to the nearest 20 mg to accommodate capsule strength.
  3. Subjects should be instructed to swallow capsules whole and in rapid succession and to not chew capsules. If vomiting occurs during the course of treatment, no re-dosing of the subject is allowed before the next scheduled dose.
  4. Temozolomide should be taken on an empty stomach. It should be administered at approximately the same time every day within and during each cycle. In general, patient tolerability is best when the drug is given at bedtime with antiemetics one hour prior to temozolomide.
  5. Since this is an oral drug, episodes of emesis will result in under dosing. Prophylactic antiemetics (oral metoclopramide is preferred, either oral or intravenous administration 5-HT3 antagonist could also be used if intolerable or not response to metoclopramide) must be administered to all subjects prior to temozolomide administration.

     7.6 Concomitant Treatments

     Concomitant medications allowed and not allowed are described below:

     Allowed:

     • Ancillary treatments will be given as medically indicated.

     • Antiemetics or antiallergic medication are permitted. Proton pump inhibitor or H2 block is permitted for prevention or treatment of steroid related peptic ulcer.

     • G-CSF is recommended for patients who have absolute neutrophil count (ANC) <500 /mm3, neutropenic fever or documented infection while neutropenic. Prophylactic use of G-CSF could be decided by treating physicians.

     • Preventive oral or i.v. antibiotics when neutropenia < 500/mm3 without fever are recommended, but the decision to use antibiotics in this case will be left to the current policy within the different hospitals.

     • Lamivudine 100 mg orally once a day is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
     * Prophylactic anticonvulsant agents are not recommended. For patients with seizure anticonvulsant agents could be used without dose adjustment of chemotherapy.

     Not Allowed:
     * The patient will not receive other investigational drugs and anticancer treatment while on study.

     7.7 Recommended Treatment for Progression or Residual Disease If patients have progression disease during treatment or residual disease after concurrent whole brain chemoradiation, further treatments will be decided by treated physician. We recommended BOMES16 regimen with or without modification for patients with suitable general condition.

  9 OFF-STUDY CRITERIA A patient will be discontinued from the study under the following circumstances

  • Disease progression beyond brain parenchyma during protocol treatment

  • Residual disease or relapse after completion of WBRT

  • Treatment schedule delay longer than 35 days

  • Patients couldn't be done any dose reduction listed in section 8.1 and 8.2.

  • Patients develop any condition of the exclusion criteria
  * Patients with poor compliance
  * Patient wishes to withdraw from this study at his/her own request

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all the following criteria to be eligible for admission for the study:

1. Histologically proven central nervous system lymphoma of brain parenchyma with or without leptomeningeal involvement.
2. No evidence of systemic lymphoma.
3. Age between 18 years and 75 years.
4. With at least one measurable lesion, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 10 mm. See Section 10.2.1 for the evaluation of measurable disease.
5. Laboratory requirements :

   * Hematology: Neutrophils≧ 1500/mm3, Hemoglobin≧ 10 g/dL, and Platelet count≧ 100000/mm3.
   * Hepatic function: Total bilirubin level≦ 1.5x upper normal limit (UNL), ALT (SGPT) and AST (SGOT)≦ 2.5 x UNL.
   * Renal function: Creatinine≦ 1.5 mg/dL.
6. No prior malignancy (excluding in situ carcinoma of the cervix or non- melanomatous skin cancer) unless disease free for at least 5 years.
7. Signed informed consent.
8. Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

Patient meets any of the following will be excluded form the study.

1. Patients who are seropositive for HIV, AIDS, use of immunosuppressant or who are post organ transplant are not eligible.
2. Previously treated with chemotherapy, radiotherapy or other investigational agents. Patients with corticosteroid use are considered eligible.
3. With ocular involvement or with any lesion beyond brain parenchyma except leptomeningeal.
4. Pregnant, or lactating patients; patients of childbearing potential must implement adequate contractive measures during study participation.
5. Other serious illness or medical conditions:

   * Congestive heart failure or unstable angina pectoris. High risk uncontrolled arrhythmias.
   * Uncontrolled infection (active serous infections that are not controlled by antibiotics.
6. Concurrent treatment with any other experimental drugs.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-11; Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Primary : To evaluate objective tumor response rate


SECONDARY OUTCOMES:
Secondary : To assess toxicity profile
To assess time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hung Lin, M.D., Principal Investigator — National Taiwan University Hospital; Ann-Lii Cheng, Ph.D., Study Chair — National Taiwan University Hospital
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei